CLINICAL TRIAL: NCT06363734
Title: Osimertinib Plus Dalpiciclib in Patients With EGFR-mutant, CDK4/6 Pathway Aberrant, Advanced Non-small Cell Lung Cancer Following Acquired Resistance on Third-generation EGFR TKI： a Single-arm Phase II Trial
Brief Title: Osimertinib Plus Dalpiciclib in Patients With EGFR-mutant, CDK4/6 Pathway Aberrant, Advanced Non-small Cell Lung Cancer Following Acquired Resistance to Third-generation EGFR TKI: a Phase II Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAL20240409
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Non-small Cell Lung Cancer; EGFR Activating Mutation; Cell Cycle Deregulation; EGFR-TKI Resistant Mutation
Keywords: NSCLC; EGFR activating mutations; Third-generation EGFR-TKI; Cell cycle signaling pathway aberrations; CDK4/6 inhibitors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; dalpiciclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- osimertinib in combination with dalpiciclib (Experimental)
  Interventions: Drug: Osimertinib plus Dalpiciclib

INTERVENTIONS:
Drug: Osimertinib plus Dalpiciclib — osimertinib 80mg daily plus dalpiciclib 125mg daily for 21 days followed by 7 days off in each 28-day treatment cycle

SUMMARY:
This study is a prospective, single-arm, phase II trial. It is aimed to evaluate the efficacy and safety of the combination of osimertinib and dalpiciclib in patients with EGFR-mutant, CDK4/6 pathway aberrant, advanced NSCLC following acquired resistance to third-generation EGFR TKI.

DETAILED DESCRIPTION:
After signing informed consents and completing the screening phase, eligible subjects who meet the enrolment criteria receive the treatment with once-daily osimertinib 80 mg plus dalpiciclib 125 mg daily for 21 consecutive days followed by 7 days off in each 28-day cycle until objective disease progression, intolerable toxicity, or other events that subjects need to be withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0 to 2 with a minimum life expectancy of 12 weeks
* Advanced non-small cell lung cancer with EGFR-sensitive mutation
* Confirmed medical history of acquired resistance to third-generation EGFR TKI
* Concurrent CDK4/6 pathway gene dysfunctional aberrations
* Evaluable or measurable disease as defined by RECIST, Version 1.1
* At least one prior line of systemic chemotherapy
* Adequate organ function

Exclusion Criteria:

* Prior treatment with any CDK4/6 inhibitor
* Active uncontrolled/unstable CNS metastases, carcinomatous meningitis, or leptomeningeal disease
* Unresolved toxicities from any prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2 prior platinum therapy related neuropathy.
* active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy (eg, ulcerative disease, uncontrolled nausea, vomiting, diarrhoea Grade ≥2, malabsorption syndrome or previous significant bowel resection).
* Unstable angina pectoris, Congestive heart failure, Acute myocardial infarction, Stroke or transient ischemic attack or other uncontrolled cardiovascular disease currently or within the last 6 months, Mean resting correct QT interval (QTcF) >470 msec for women and >450 msec for men at Screening, obtained from 3 ECGs using the screening clinic ECG machine derived QTcF value.
* Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy.
* Major surgical procedures ≤28 days of beginning study drug or minor surgical procedures ≤7 days
* Evidence of severe or uncontrolled systemic diseases, including renal transplant, active bleeding diatheses or uncontrolled hypertension
* Active hepatitis B or C or known serious active infection e.g. tuberculosis or human immunodeficiency virus. Viral testing is not required for assessment of eligibility for the study.
* Known serious active infection including, but not limited to, tuberculosis, or human immunodeficiency virus (positive human immunodeficiency virus 1/2 antibodies).
* Presence of other active cancers, or history of treatment for invasive cancer, within the last 5 years.
* Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 2 weeks prior to start of study treatment.
* Past medical history of interstitial lung disease(ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
* History of liver cirrhosis of any origin and clinical stage; or history of other serious liver disease or chronic disease with relevant liver involvement, with or without normal LFTs,
* Any cytotoxic chemotherapy, investigational agents or other anticancer drugs for the treatment of advanced NSCLC from a previous treatment regimen or clinical study within 14 days prior to the first dose of study treatment with the exception of monotherapy osimertinib which may continue uninterrupted during screening.
* Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers or inhibitors of CYP3A4 within 3 weeks of the first dose of study treatment
* Participation in another clinical study with a cytotoxic, investigational product (IP), or other anticancer drug for the treatment of advanced NSCLC if received IP from that study within 14 days of the first dose of study treatment.
* Known hypersensitivity to the active or inactive excipients of osimertinib or dalpiciclib or drugs with a similar chemical structure or class.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 12 months

SECONDARY OUTCOMES:
disease control rate (DCR) | 12 months
Duration of Response (DoR) | 12 months
Progression Free Survival (PFS) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic Medical Oncology, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided